CLINICAL TRIAL: NCT01532050
Title: PROMAD : Predicting Therapeutic Outcome of Mandibular Advancement Device Treatment in Obstructive Sleep Apnea
Brief Title: PROMAD: Predicting Therapeutic Outcome of Mandibular Advancement Device Treatment in Obstructive Sleep Apnea
Acronym: PROMAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ethisch.comite@uza.be (Other)
Responsible Party: Sponsor-Investigator, ethisch.comite@uza.be, prof. Marc Braem, DDS, PhD, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IWT MRA UZA
Record Dates: First submitted 2012-01-30; First posted 2012-02-13 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSAS; American Academy of Sleep Medicine Task Force
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mandibular Advancement Device (MAD) (Other): Mandibular Advancement Device (MAD)
  Interventions: Device: Mandibular Advancement Device ( MAD)

INTERVENTIONS:
Device: Mandibular Advancement Device ( MAD)

SUMMARY:
The present research intends to focus clinically on selecting the right type of patient for mandibular advancement devices (MAD) therapy using screening tools such as advanced imaging and computational methods based on CT-Scan images as well as drug-induced sleep nasendoscopy techniques with simulation of the mandibular repositioning. The core of the research project relies on known and established methods accepted in several neighboring fields, but aims at the transfer of this knowledge by integrating it into this new domain. Doing so, the proposed biomedical research is directed towards clinical applications that incorporate innovative developments on the level of the diagnosis and therapy of a specific disease, being obstructive sleep apnea syndrome (OSAS). Furthermore, this study aims at registering objective compliance during MAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* body mass index (BMI) ≤ 35 kg/m²
* OSAS, as defined by the American Academy of Sleep Medicine Task Force
* apnea-hypopnea index (AHI) < 50

Exclusion Criteria:

* Other sleep disorders (i.e. parasomnias)
* Invasive upper airway surgery for sleep-disordered breathing
* Known genetic disorders with craniofacial and/or upper airway malformations
* Use of benzodiazepine and/or antidepressants
* Known history of psychiatric disease
* Known history of fibromyalgia and/or chronic fatigue syndrome
* Dental contra-indications: functional restrictions of the temporomandibular joint, insufficient dentition with pathological changes, insufficient retention for MAD use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Predictive value of DISE and CFD | 3 months
  Positive and negative predictive values for AHI based treatment outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Van Gaver H, Op de Beeck S, Dieltjens M, De Backer J, Verbraecken J, De Backer WA, Van de Heyning PH, Braem MJ, Vanderveken OM. Functional imaging improves patient selection for mandibular advancement device treatment outcome in sleep-disordered breathing: a prospective study. J Clin Sleep Med. 2022 Mar 1;18(3):739-750. doi: 10.5664/jcsm.9694. PMID 34608859
- [Derived] Op de Beeck S, Dieltjens M, Azarbarzin A, Willemen M, Verbraecken J, Braem MJ, Wellman A, Sands SA, Vanderveken OM. Mandibular Advancement Device Treatment Efficacy Is Associated with Polysomnographic Endotypes. Ann Am Thorac Soc. 2021 Mar;18(3):511-518. doi: 10.1513/AnnalsATS.202003-220OC. PMID 32946702
- [Derived] Van de Perck E, Op de Beeck S, Dieltjens M, Vroegop AV, Verbruggen AE, Willemen M, Verbraecken J, Van de Heyning PH, Braem MJ, Vanderveken OM. The relationship between specific nasopharyngoscopic features and treatment deterioration with mandibular advancement devices: a prospective study. J Clin Sleep Med. 2020 Jul 15;16(7):1189-1198. doi: 10.5664/jcsm.8474. PMID 32267227
- [Derived] Op de Beeck S, Dieltjens M, Verbruggen AE, Vroegop AV, Wouters K, Hamans E, Willemen M, Verbraecken J, De Backer WA, Van de Heyning PH, Braem MJ, Vanderveken OM. Phenotypic Labelling Using Drug-Induced Sleep Endoscopy Improves Patient Selection for Mandibular Advancement Device Outcome: A Prospective Study. J Clin Sleep Med. 2019 Aug 15;15(8):1089-1099. doi: 10.5664/jcsm.7796. PMID 31482830
- [Derived] Dieltjens M, Verbruggen AE, Braem MJ, Wouters K, Verbraecken JA, De Backer WA, Hamans E, Van de Heyning PH, Vanderveken OM. Determinants of Objective Compliance During Oral Appliance Therapy in Patients With Sleep-Disordered Breathing: A Prospective Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Oct;141(10):894-900. doi: 10.1001/jamaoto.2015.1756. PMID 26402736